CLINICAL TRIAL: NCT02692001
Title: A Randomized Controlled Trial to Evaluate the Impact of Child Friendly Menu Labelling Designs on Food Choices by Parents and Children in an Inpatient Hospital Setting
Brief Title: Child Friendly Menu Labelling and Food Choices
Acronym: MealTrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Staff Physician , Division of Endocrinology, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1000048168
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current MealTrain menu (No Intervention): This is the current menu being employed for food ordering in the pediatric inpatient wards.
- Intervention MealTrain menu (Experimental): The intervention menu included child-friendly labeling (attractive characters, fun food names and traffic light system) to encourage healthier choices.
  Interventions: Other: Intervention MealTrain menu

INTERVENTIONS:
Other: Intervention MealTrain menu — Nutrition education was incorporated using an interpretive traffic light system menu labeling. Dietitians categorized current menu items as green, yellow and red based on fiber, added sugar, saturated fats, and sodium content. A section entitled "Eat like a superhero" was created to prime children to consider what their potential role models choose, and incorporates descriptive names, suggest sample breakfast, lunch and dinner meals with photographs of portion sizes. Original cartoon female grapes and male broccoli superhero characters were created to employ promotional techniques specifically to promote fruits and vegetable selection for boys and girls.
  Arms: Intervention MealTrain menu

SUMMARY:
Childhood obesity is a major problem in Canada. Children are eating larger portions and have easier access to high-fat, high-sugar foods and drinks. Menu labelling is a promising tool to teach families about healthier choices. The investigators will study the impact of combining child-friendly superhero food labels, fun food names, and a traffic light system on the food choices of children and their parents at SickKids. The investigators will use the hospital inpatient food ordering system (Meal Train) and look at food orders and eating patterns before and after introduction of the revised Meal Train menu. Only the design format of the menu was changed and all menu items remained unchanged. The investigators will also survey the families on their thoughts about the menu. This study will help doctors and dietitians develop strategies to deliver nutrition education to families.

DETAILED DESCRIPTION:
Childhood obesity is recognized as a major public health epidemic in Canada with over 31.5% of all 5- to 17-year-olds being overweight or obese. The etiology of this increase in childhood obesity can be attributed to trends in children's diets that include increasing access to foods high in fats, added sugars, and eating outside the home with routine exposure to large portions of energy-dense, nutrient-poor foods. Menu labelling and point-of-purchase nutrition information is a promising potential cost effective public health strategy and utilized in the adult population. In this study, the investigators plan to evaluate the impact of a combination of labelling techniques including attractive characters, descriptive food names and traffic light system on food choices made by children and their parents in an inpatient hospital setting at the Hospital for Sick Children. The investigators will assess patient ordering and consumption patterns before and after the introduction of a revised educational Meal Train menu. A crossover randomized control trial design will be employed to identify changes in fruit and vegetable intake, healthy ("green light") option intake, number of sweetened beverages and energy-dense nutrient-poor ("red light") foods chosen as well as the number of children that meet the Canadian Food Guide (CFG) daily serving recommendations. As a secondary analysis, the investigators will be collecting participant's age, sex and weight-for-age z-score (as defined by the World Health Organization guidelines) to investigate any potential relationships between these variables and food ordering patterns before and after introduction of the proposed educational menu. A questionnaire will also be distributed to assess parent and child perceptions of the revised Meal Train menu. The investigators hypothesize patient ordering and consumption patterns before and after the introduction of a revised educational Meal Train menu will promote healthier food selections. While this type of intervention has been studied in hypothetical restaurants and cafeteria setting, this will be the first study conducted in a hospital setting with pediatric inpatients and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a general pediatrics or subspecialty wards
* Fluent in written English

Exclusion Criteria:

* NPO or receiving parenteral nutrition at any point in their admission
* Specialized diet e.g. celiac, purée, renal diet, or high energy diet
* Those exposed to educational intervention menu in first 2 weeks who remain on ward following the crossover period

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 163 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Evaluate patient ordering patterns before and after the introduction of the revised educational Meal Train menu. | 1 month
  Specifically, the investigators will determine whether the revised Meal Train menu results in:
  1. Increased fruit and vegetable ordered
  2. A decrease in the number of sweetened beverages and energy-dense nutrient-poor ("red light") foods ordered
  3. A higher number of individual daily food orders that meet the Canadian Food Guide (CFG) daily serving recommendations.
  4. An increase in healthy foods ordered (green light options)

SECONDARY OUTCOMES:
Relationship between patient demographics and meal orders | 1 month
  The relationship between age, sex and weight-for-age z-score (as defined by the World Health Organization guidelines) and food ordering/consumption patterns before and after introduction of the proposed educational menu
Impact of child-friendly menu designs on food orders | 1 month
  Foods highlighted by specific aspects of the menu (attractive characters and descriptive food names OR traffic light system) and whether their presence impacted food ordering patterns.
Evaluation of meal consumption | 1 month
  Meal consumption: Meal trays of 20% of orders ( 2 days/study period) will be collected and leftover food measured by volunteer dietetic interns.
  Consumption patterns will be evaluated before and after the introduction of the revised educational Meal Train menu. Specifically, we will determine whether the revised Meal Train menu results in:
  Specifically, we will determine whether the revised Meal Train menu results in:
  1. Increased fruit and vegetable consumed
  2. A decrease in the number of sweetened beverages and energy-dense nutrient-poor ("red light") foods consumed
  3. A higher number of individual daily food consumption that meet the Canadian Food Guide (CFG) daily serving recommendations.
  4. An increase in healthy foods consumed (green light options)
Parent/child perceptions of the revised Meal Train menu | 1 month
  Survey: a one page paper survey for both parent and child (age > 10) to assess perceptions of menu labelling on food ordering

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish in a peer reviewed journal, as well as presnt at national and international conferences (Canadian Pediatric Endocrine Group, International Conference for Obesity and Canadian Pediatric Society )

REFERENCES:
- [Derived] Basak S, Steinberg A, Campbell A, Dupuis A, Chen S, Dayan AB, Dello S, Hamilton J. All Aboard Meal Train: Can Child-Friendly Menu Labeling Promote Healthier Choices in Hospitals? J Pediatr. 2019 Jan;204:59-65.e3. doi: 10.1016/j.jpeds.2018.08.073. Epub 2018 Sep 28. PMID 30274925